CLINICAL TRIAL: NCT04064476
Title: The Effect of Long-acting Antipsychotic on Schizophrenia Patients With Violence Risk : a Observational Cohort Study
Brief Title: The Effect of Long-acting Antipsychotics on Schizophrenia Patients With Violence Risk
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yi Li MD, PhD, Professor, Huazhong University of Science and Technology
Other Study IDs: WG17A002II
Record Dates: First submitted 2019-07-25; First posted 2019-08-22 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia; violence risk; long-acting antipsychotics
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Will take blood sample and kept it for further analysis after get agreement from the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Paliperidone Palmitate — This is a observational study, to see the effect of paliperidone palmitate on schizophrenia patient with violence risk. The intervention is determined by clinical practice in real world setting, only schizophrenia patient with violence risk and treated with Paliperidone Palmitate will be invited to join the observational study.

SUMMARY:
This is a 49 weeks prospective, non-interventional cohort study. To observe the effect of long-acting injection antipsychotic(LAI), paliperidone palmitate on prevention of recurrence and symptom control in schizophrenia patients with violence risk. This study can be extended according to the implementation of the project and extended follow-up time.

DETAILED DESCRIPTION:
This is a 49 weeks prospective, observational cohort study. Wuhan initiated a project to improve the LAI treatment in schizophrenia patient with violence risk. This observational study will build the cohort of schizophrenia patient with violence risk and treated with LAI paliperidone palmitate. The effect of long-acting antipsychotic, paliperidone palmitate, will be observed on prevention of recurrence and symptom control in these patients. safety information and laboratory tests result will also be collected. This study can be extended according to the implementation of the project and extended follow-up time.

ELIGIBILITY:
Patient who has violence risk and in the supervise of government system, and treated with paliperidone palmitate will be invited to the observational study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient who has violence risk and in the supervise of government system, and treated with paliperidone palmitate, and signed the informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2019-08-18 (Actual); Primary Completion 2021-08-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale(PANSS) | 49 Weeks
  PANSS score change. PANSS was used to assess schizophrenia psychopathology symptoms of subjects. PANSS gave a total score (total score of 30 items) and three subscale scores, positive subscale (7 items), negative subscale (7 items), general psychopathology symptoms subscale (16 items) . Each scale rated from 1 (none) to 7 (very heavy).

SECONDARY OUTCOMES:
Modified Overt Aggression Scale (MOAS) | 49 Weeks
  Score change of Modified Overt Aggression Scale (MOAS ). MOAS is used to assess aggressive behavior of psychosis patients. Including Verbal aggressive, aggressive to property, aggressive to self, aggressive to others, and total score. Each domain with score 0 to 4, total weighted score 0 to 40
Violence Risk Assessment For Psychiatric Patients | 49 Weeks
  The Violence risk assessment scale for psychotic patients is a 0-5 score scale, established by the China national working group and used in the China National Continuing Management and Intervention Program for Psychoses, to evaluate psychotic patients' risk of violence [12]. 0 is no violence. 1 is verbal threat, shouting, but without aggressive behavior. 2 is beating or smashing property, limited in home. 3 is beating or smashing property in any place, cannot be dissuaded, but did not hurt people. 4. Consistently beating or smashing property or people in any place, cannot be dissuaded. 5, Any violent behavior with the dangerous weapon, or arson.
Hospitalization frequency | 49 Weeks
  Hospitalization due to schizophrenia during 49 weeks
WHO Quality of Life-BREF (WHOQOL-BREF) of patients | 49 Weeks
  The patients' WHOQOL-BREF score. The WHOQOL-BREF offers a short, generic, subjective quality of life (QoL) measure, 26 important questions are scored in environmental, social, physical and psychological domains, each question from 1-5.
Visual Analogue Scale-100 (VAS 100) of caregiver treatment satisfaction | 49 Weeks
  The Caregiver' VAS 100 score change. caregiver rate according to their treatment satisfaction, score from 1( extremely unsatisfied) to 100( extremely satisfied. measure, 26 important questions are scored in environmental, social, physical and psychological domains, each question from 1-5
Visual Analogue Scale-100 (VAS 100) of patients treatment satisfaction | 49 Weeks
  The patients' VAS 100 score change. Patients rate according to their treatment satisfaction, score from 1( extremely unsatisfied) to 100( extremely satisfied.
Visual Analogue Scale-100 (VAS 100) of caregiver's treatment satisfication | 49 Weeks
  The caregivers' VAS 100 score change.Caregivers rate according to their treatment satisfication, score from
  1( extremely unsatisfied) to 100( extremely satisfied.
Personal and Social Performance Scale (PSP) | 49 Weeks
  PSP was a clinical scoring tool that was used for personal and social function assessment in schizophrenia subjects, and the score ranged between 1 and 100. The scale defined a continuous functional status, from overall function impaired (completely lack of independent basic functions, survival is significantly dangerous) to function well. The scale takes four functional dimensions into account: a) social useful activities, including work and study, b) the relationship between the individual and society, c) self-care, and d) disturbing and aggression
Treatment Emergent Symptom Scale (TESS) | 49 Weeks
  Treatment Emergent Symptom Scale (TESS) is a checklist including common adverse event in psychotic treatment.
  each item rate from 0( no) to 4 (heavy)
Electrocardiogram (ECG) | 49 Weeks
  ECG testing should be performed in a quiet non-interference (such as TV, mobile) environment for the subjects. Before testing ECG the subjects should rest in the supine position for at least 5 minutes and should be limited to conversation or physical activity. Twelve-lead ECG was recorded by 25 mm/sec paper speed, measuring RR, PR, QRS and QT intervals
Adverse events | 49 Weeks
  The frequency of adverse events in the treatment period
Calgary Depression Scale of Schizophrenia(CDSS) | 49 weeks
  Calgary Depression Scale of Schizophrenia is a scale to assess the depression symptom in schizophrenia patients, It comprises of 9 items, each item has 4 grade(0, 1, 2, 3), the higher score means more serious depression. Maximize score is 27 points. Above 6 points reflect has depression symptom.
Liver function tests | 49 weeks
  Liver function tests are groups of blood tests that provide information about the state of a patient's liver. In this case includes alanine transaminase (ALT) and aspartate transaminase (AST).
Renal function tests | 49 weeks
  Renal function tests includes blood tests that provide information about blood urea nitrogen (BUN) and creatinine.
Blood glucose tests | 49 weeks
  Using blood glucose monitoring to perform fingerprick type of glucose meter.
Blood lipid tests | 49 weeks
  Liver function tests are groups of blood tests that provide information about high density lipoprotein (HDL), low density lipoprotein (LDL) and triglyceride.
STROOP test | 49 weeks
  The test is considered to measure selective attention, cognitive flexibility and processing speed, and it is used as a tool in the evaluation of executive functions. The color of the character should be named both in undisturbed and disturbed condition. The time spent in both cases will be compared
RBANS | 49 weeks
  Repeatable Battery for the Assessment of Neuro-psychological Status (RBANS), The RBANS provides SS based on same-aged peers for 5 indexes of neuropsychological functioning: Attention, Language, Visuospatial-Construction, Immediate Memory, and Delayed Memory . These indexes combine to compute a total scale score of cognitive functioning
Interpersonal Reactivity Index(IRI) | 49 weeks
  Interpersonal Reactivity Index. The IRI was designed to assess empathy.It contains 4 sub-scales, each with 7 items. It uses a 5-item Likert scale with two anchors (A = Does not describe me well; E= Describes me very well). Responses can be averaged (using 0 to 4 or 1 to 5 endpoints) or summed (using 0 to 28 or 7 to 35 ranges). The IRI is a continuous measure of empathy in normal populations and not a categorical ,measure ("high empathy" versus "low empathy").
Facial Emotion Recognition scale | 49 weeks
  Computer-morphed images derived from the facial features of real individuals, each showing a specific emotion, are displayed on the screen, one at a time. Each face is displayed for 200ms and then immediately covered up to prevent residual processing of the image. The participant must select which emotion the face displayed from 6 options (sadness, happiness, fear, anger, disgust or surprise). The outcome measures for ERT cover percentages and numbers correct or incorrect and overall response latencies, which can be looked at either across individual emotions or across all emotions at once.
Toronto Alexithymia Scale(TAS) | 49 weeks
  Toronto Alexithymia Scale, the TAS is a 20-item instrument that commonly used measures of alexithymia. It is a self-report scale that is comprised of 20 items. Items are rated using a 5-point Likert scale whereby 1 = strongly disagree and 5 = strongly agree. There are 5 items that are negatively keyed (items 4, 5, 10, 18 and 19). The total alexithymia score is the sum of responses to all 20 items, while the score for each subscale factor is the sum of the responses to that subscale. The TAS-20 uses cutoff scoring: equal to or less than 51 = non-alexithymia, equal to or greater than 61 = alexithymia. Scores of 52 to 60 = possible alexithymia.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Li, Dorctor, Principal Investigator — HuaZhong university, Wuhan mental health center
Locations (1):
- Wuhan mental health center, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
No share plan